CLINICAL TRIAL: NCT04031703
Title: Study Comparing Paclitaxel Plus Carboplatin Versus Anthracyclines Followed by Docetaxel as Adjuvant Chemotherapy for Triple Negative Breast Cancer
Brief Title: Study Comparing Paclitaxel Plus Carboplatin Versus Anthracyclines Followed by Docetaxel as Adjuvant Chemotherapy for Triple Negative Breast Cancer (PATTERN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATTERN
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Epirubicin; Cyclophosphamide; Fluorouracil; Docetaxel

STUDY DESIGN:
Intervention Model Description: Arm 1：6 cycles of PC (Paclitaxel 80 mg/m2 ivgtt d1,8,15+ Carboplatin Auc = 2 ivgtt d1,8,15, 28 days per cycle).
  Arm 2：3 cycles of FEC (epirubicin100 mg/m2 ivgtt d1+Cyclophosphamide 500 mg/m2 iv d1+ 5-fluorouracil 500 mg/m2 iv d1, 21 days per cycle) followed by 3 cycles of Docetaxel (Docetaxel 100mg/m2, ivgtt d1, 21 days per cycle)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6 cycles of PC adjuvant chemotherapy (Experimental): 6 cycles of PC (Paclitaxel 80 mg/m2 ivgtt d1,8,15+ Carboplatin Auc = 2 ivgtt d1,8,15, 28 days per cycle).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- 3 cycles of FEC followed by 3 cycles of Docetaxel (Active Comparator): 3 cycles of FEC (epirubicin100 mg/m2 ivgtt d1+Cyclophosphamide 500 mg/m2 iv d1+ 5-fluorouracil 500 mg/m2 iv d1, 21 days per cycle) followed by 3 cycles of Docetaxel (Docetaxel 100mg/m2, ivgtt d1, 21 days per cycle)
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: 5-fluorouracil; Drug: Docetaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel chemotherapy (injection)
  Arms: 6 cycles of PC adjuvant chemotherapy
Drug: Carboplatin — Carboplatin chemotherapy (injection)
  Arms: 6 cycles of PC adjuvant chemotherapy
Drug: Epirubicin — Epirubicin chemotherapy (injection)
  Arms: 3 cycles of FEC followed by 3 cycles of Docetaxel
Drug: Cyclophosphamide — Cyclophosphamide chemotherapy (injection)
  Arms: 3 cycles of FEC followed by 3 cycles of Docetaxel
Drug: 5-fluorouracil — 5-fluorouracil chemotherapy (injection)
  Arms: 3 cycles of FEC followed by 3 cycles of Docetaxel
Drug: Docetaxel — Docetaxel chemotherapy (injection)
  Arms: 3 cycles of FEC followed by 3 cycles of Docetaxel

SUMMARY:
This is a prospective, multisite, randomized, open-lable Phase III clinical trial (PATTERN study) comparing Paclitaxel Plus Carboplatin versus Anthracyclines followed by docetaxel as adjuvant chemotherapy for triple negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-65 years old;
2. Patient has localized invasive breast carcinoma, and is ER-/PR-/HER2- confirmed by histopathology after early breast cancer surgery（HER2-negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH), or Silver in situ hybridization (SISH)) test is required by local laboratory testing.), positive lymph node or negative lymph node with at least one of the following conditions: (1) histological grade II or III; (2) tumor size > 0.5
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN，and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
5. Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy）;
2. Has bilateral breast cancer;
3. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastic (Stage 4) breast cancer;
5. Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
6. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
7. Patients participating in other clinical trials at the same time;
8. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
9. Has known allergy to taxane and excipients.
10. Has severe or uncontrolled infection;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 year

SECONDARY OUTCOMES:
distant metastasis free survival | 5 year
event free survival | 5 year
overall survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University